CLINICAL TRIAL: NCT03480308
Title: Effect of Addition of Fentanyl or Dexamethasone or Both to Bupivacaine in Paravertebral Block for Patients Undergoing Major Breast Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amonios khalil, doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: paravertebral block
Record Dates: First submitted 2018-03-16; First posted 2018-03-29 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Paravertebral Block
MeSH Terms: interventions — Fentanyl; Dexamethasone; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Patients will receive ultrasound guided paravertebral block and stratified into 3 groups according to medication used :
  Group 1 : bupivacaine (0.5%) 20 ml , fentanyl 1 μg/kg Group 2 : bupivacaine (0.5%) 20 ml , dexamethasone 4 mg Group 2 : bupivacaine (0.5%) 20 ml , fentanyl 1 μg/kg , dexamethasone 4 mg
Who Masked: Investigator
Masking Description: Randomization Will be Done Using Computer Generated Tables
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bupivacaine fentanyl group (Active Comparator): Patients will receive bupivacaine (0.5%) 20 ml , fentanyl 1 μg/kg in paravertebral block
  Interventions: Drug: Fentanyl; Drug: Bupivacaine
- Bupivacaine dexamethasone group (Active Comparator): Patients will receive bupivacaine (0.5%) 20 ml , dexamethasone 4 mg in paravertebral block
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine
- Bupivacaine fentanyl dexamethasone group (Active Comparator): Patients will receive bupivacaine (0.5%) 20 ml , fentanyl 1 μg/kg , dexamethasone 4 mg in paravertebral block
  Interventions: Drug: Fentanyl; Drug: Dexamethasone; Drug: Bupivacaine

INTERVENTIONS:
Drug: Fentanyl — Patients will receive bupivacaine (0.5%) 20 ml , fentanyl 1 μg/kg in paravertebral block
  Arms: Bupivacaine fentanyl dexamethasone group; Bupivacaine fentanyl group
Drug: Dexamethasone — Patients will receive bupivacaine (0.5%) 20 ml , Dexamethasone 4mg in paravertebral block
  Arms: Bupivacaine dexamethasone group; Bupivacaine fentanyl dexamethasone group
Drug: Bupivacaine — Bupivacaine

SUMMARY:
This study evaluated the analgesic efficacy of fentanyl and dexamethasone in combination with bupivacaine for single-shot paravertebral block (PVB) in patients undergoing major breast surgery.

DETAILED DESCRIPTION:
This study evaluated the analgesic efficacy of fentanyl and dexamethasone in combination with bupivacaine for single-shot paravertebral block (PVB) in patients undergoing major breast surgery.

Patients will receive ultrasound guided paravertebral block and stratified into 3 groups according to medication used :

Group 1 : bupivacaine (0.5%) 20 ml , fentanyl 1 μg/kg Group 2 : bupivacaine (0.5%) 20 ml , dexamethasone 4 mg Group 2 : bupivacaine (0.5%) 20 ml , fentanyl 1 μg/kg , dexamethasone 4 mg

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years.
* Sex: females
* ASA physical status: I-II.
* Operation: major breast surgery

Exclusion Criteria:

* - Patient refusal.
* History of cardiac disease, psychological disorders, respiratory diseases including asthma, renal or hepatic failure.
* Coagulation disorders.
* Infection at the puncture site
* Allergy to study medications.
* Chronic use of pain medications.
* Respiratory tract in¬fection within the last 2 weeks.
* Neurological deficit

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Time to first analgesic request | one day postoperative
pain assessment | one day postoperatively
  Pain assessment by the aid of Visual analogue scale (VAS) Ranging from 0=no pain, 10=excruciating pain higher values represent worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Amonios khalil, Study Director — Faculty of medicine-Assiut university-Egypt
Locations (1):
- Amonios Khalil gerges, Asyut, Egypt